CLINICAL TRIAL: NCT01221142
Title: Pilot Study of Hypothermia for Intracerebral Hemorrhage in Croatia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Rijeka (Other)
Collaborators: PharmamedMado d.o.o., Zagreb, Croatia (Unknown)
Responsible Party: University Hospital Rijeka, Igor Antončić MD
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HfICHiC
Record Dates: First submitted 2010-10-13; First posted 2010-10-14 (Estimated); Last update posted 2010-12-28 (Estimated); Status verified 2010-10

CONDITIONS: Hypothermia; Primary Intracerebral Hemorrhage; Signs and Symptoms
Keywords: Hypothermia, ICH
MeSH Terms: conditions — Hypothermia; Signs and Symptoms; Hepatitis, Infectious Canine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hypothermia (Experimental): Device: Cincinnati Sub-Zero Hyper-Hypothermia to core temperature of 34C for 24 hours, rewarming rate 0,5/2h until the patient reaches 36,5C
  Interventions: Device: Cincinnati Sub-Zero," Blanketrol III"

INTERVENTIONS:
Device: Cincinnati Sub-Zero," Blanketrol III"

SUMMARY:
In this pilot study the researchers will investigate efficacy of hypothermia in the early stage of treatment patients with primary intracerebral hemorrhage.

DETAILED DESCRIPTION:
The purpose of this pilot trial is to determine whether hypothermia improves neurological outcome (measured as 3 and 6 months after the onset of symptoms using mRS, GOS and BI) in patients who has suffered a primary intracerebral hemorrhage. The patients with primary intracerebral hemorrhage presented with coma (GCS ≤ 8) and ICH score 2-4 will be included. Induction of hypothermia will be initiated within 6 hours of symptoms onset. Patients will be cooled to core temperature of 34°C during 24 hours using non-invasive temperature management (Cincinnati Sub-Zero). The temperature will be measured continuously by esophageal system. After 24 hours of successful cooling, the target temperature will be gradually raised to achieve slow re-warming of 0.5°C / 2 h until the core temperature reaches 36,5°C.

During hypothermia ECG, blood pressure, oxygen saturation and intracranial pressure will be measured continuously and registered every 30 min. The first CT scan of the brain, after initial, will be done early after normothermia is reached.

ELIGIBILITY:
Inclusion Criteria:

* GCS ≤ 8
* ICH score 2-4
* symptom onset within 6 hours
* ages 18 - 80

Exclusion Criteria:

* pregnancy
* hemodynamical unstability
* recent myocardial infarction
* systolic blood pressure < 90 mm Hg

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2011-01; Primary Completion 2011-09; Study Completion 2012-06

PRIMARY OUTCOMES:
Neurological outcome | 3 months after the onset
Neurological outcome | 6 months after the onset

SECONDARY OUTCOMES:
Mortality | 1 week
Mortality | 1 month
Mortality | 6 months
The incidence of significant cardiac arrhythmias, infections, severe disturbances of electrolytes | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Igor Antoncic, MD, MSc, Principal Investigator — Intensive Care Unit, Departmen of Neurology, University Hospital Rijeka, Croatis
Locations (1):
- Intensive Care Unit, Department of Neurology, University Hospital Rijeka, Rijeka, Croatia